CLINICAL TRIAL: NCT03966911
Title: Performance Evaluation of an Advanced Algorithm With CGM in Adults, Adolescents, and Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP324
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Type 1 Diabetes Mellitus; Type2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subjects with diabetes wearing Guardian™ Sensor (3) (Other): Subjects wear Guardian™ Sensor (3) and Guardian™ Connect Transmitter over 7 days and participate in FSTs. Zero calibration sensor algorithm applied to raw sensor data.
  Interventions: Device: Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter

INTERVENTIONS:
Device: Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter — Continuous Glucose Monitoring and frequent sample testing

SUMMARY:
The purpose of this study is to demonstrate the performance of the Guardian™ Sensor (3) with an advanced algorithm in subjects age 2 - 80 years, for the span of 170 hours (7 days).

DETAILED DESCRIPTION:
The study is a multi-center, prospective, single-sample correlational design without controls. The purpose of this study is to demonstrate the performance of the Guardian™ Sensor (3) with an advanced algorithm in subjects age 2 - 80 years, for the span of 170 hours (7 days).

ELIGIBILITY:
Inclusion Criteria:

1. Individual is 2 - 80 years of age at time of enrollment
2. A clinical diagnosis of type 1 or 2 diabetes for a minimum of 6 months duration as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Adequate venous access as assessed by investigator or appropriate staff
4. Subjects participating in the high and low glucose challenges must have an insulin carbohydrate ratio(s) and insulin sensitivity ratio. Subjects without ratios may participate under observation only

Exclusion Criteria:

1. Subject will not tolerate tape adhesive in the area of Guardian™ Sensor (3) placement as assessed by a qualified individual.
2. Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
4. Subject is female and has a positive pregnancy screening test
5. Female of child bearing age and who is sexually active should be excluded if she is not using a form of contraception deemed reliable by investigator
6. Subject is female and plans to become pregnant during the course of the study
7. Subject has had a hypoglycemic seizure within the past 6 months prior to enrollment
8. Subject has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to enrollment.
9. Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to enrollment.
10. Subject has a history of a seizure disorder
11. Subject has central nervous system or cardiac disorder resulting in syncope
12. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
13. Subject has a hematocrit (Hct) lower than the normal reference range (please note that patients may use prior blood draw from routine care as long as done within 6 months of screening and report of lab placed with subject source documents)
14. Subject has a history of adrenal insufficiency
15. Subject is a member of the research staff involved with the study.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - AMCR Institue, Escondido, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - SoCal Diabetes, Torrance, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center - Adults, Aurora, Colorado
  - Barbara Davis Center for Childhood Diabetes (Pediatric), Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - IDERC, Des Moines, Iowa
  - Mayo Clinic (Rochester MN), Rochester, Minnesota
  - AM Diabetes & Endocrinology Center, Bartlett, Tennessee
  - Texas Diabetes and Endocrinology, Austin, Texas
  - University of Virgina, Charlottesville, Virginia
  - Rainer Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 335 subjects (188 adult subjects and 147 pediatric subjects) consented and enrolled in the overall study. Of them, 311 subjects (169 adult subjects and 142 pediatric subjects) were eligible.
Groups:
- Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3): Adult subjects (age 18-80) wear Guardian™ Sensor (3) over 7 days and participate in FSTs.
  Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter: Continuous Glucose Monitoring and frequent sample testing
- Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3): Pediatric subjects (age 2-17) wear Guardian™ Sensor (3) over 7 days and participate in FSTs.
  Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter: Continuous Glucose Monitoring and frequent sample testing
Period: Overall Study
Arm/Group | Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) | Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3)
Started | 169 | 142
Completed | 160 | 126
Not Completed | 9 | 16
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Unable to complete study visits due to COVID-19 | 0 | 13

BASELINE CHARACTERISTICS:
Population: Demographics and other baseline characteristics were documented for eligible subjects (i.e., subjects who passed screening).
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) | Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3) | Total
Number analyzed (Participants) | 169 | 142 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (17.8) | 10.9 (4.0) | 29.9 (22.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 59 | 150
  Male | 78 | 83 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 17 | 38
  Not Hispanic or Latino | 148 | 125 | 273
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 169 | 142 | 311

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Readings Within 20% Agreement
Description: Mean of daily percentage of sensor values within 20% of Yellow Springs Instrument (YSI™*) reference value (within 20 mg/dL if sensor values < 80 mg/dL), across all participants and all Frequent Sample Testing (FST) days. Note Self-Monitoring Blood Glucose (SMBG) was used for age 2-6, instead of YSI.
Time Frame: 7 days (170 hours)
Population: Subjects with at least 1 sensor-YSI (or sensor-SMBG for subjects 2-6 years) paired point during the sensor wear
Measure: Mean (91.8% Confidence Interval); unit: Percentage of Readings
Groups:
- Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) on the Arm: Adult subjects (age 18-80) wear Guardian™ Sensor (3) on the arm over 7 days and participate in FSTs. Zero calibration sensor algorithm applied to raw sensor data.
  Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter: Continuous Glucose Monitoring and frequent sample testing
- Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) on the Abdomen: Adult subjects (age 18-80) wear Guardian™ Sensor (3) on the abdomen over 7 days and participate in FSTs. Zero calibration sensor algorithm applied to raw sensor data.
  Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter: Continuous Glucose Monitoring and frequent sample testing
- Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3) on the Arm: Pediatric subjects (age 2-17) wear Guardian™ Sensor (3) on the arm over 7 days and participate in FSTs. Zero calibration sensor algorithm applied to raw sensor data.
  Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter: Continuous Glucose Monitoring and frequent sample testing
- Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3) on the Buttock: Pediatric subjects (age 2-17) wear Guardian™ Sensor (3) on the buttock over 7 days and participate in FSTs. Zero calibration sensor algorithm applied to raw sensor data.
  Guardian™ Sensor (3) connected to a Guardian™ Connect Transmitter: Continuous Glucose Monitoring and frequent sample testing
Arm/Group | Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) on the Arm | Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) on the Abdomen | Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3) on the Arm | Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3) on the Buttock
Number analyzed (Participants) | 169 | 169 | 142 | 142
Percentage of Readings | 88.00 [86.05 to 89.95] | 87.96 [86.13 to 89.80] | 84.59 [82.02 to 87.17] | 81.05 [77.58 to 84.53]
Statistical Analysis 1: Comparison: Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) on the Arm; Test type: Superiority; p < 0.041, ANCOVA; A generalized estimating equation model was used, considering correlation structure of day of sensor wear (1-7); Intercept from ANCOVA as agreement rate = 88.00, 91.8% CI 2-sided [86.05 to 89.95] — A group sequential study design was utilized to perform interim analysis. For the final stage, the p-value is 0.041
Statistical Analysis 2: Comparison: Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) on the Abdomen; Test type: Superiority; p < 0.041, ANCOVA; A generalized estimating equation model was used, considering correlation structure of day of sensor wear (1-7); Intercept from ANCOVA as agreement rate = 87.96, 91.8% CI 2-sided [86.13 to 89.80] — A group sequential study design was utilized to perform interim analysis. For the final stage, the p-value is 0.041
Statistical Analysis 3: Comparison: Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3) on the Arm; Test type: Superiority; p = 0.041, ANCOVA; A generalized estimating equation model was used, considering correlation structure of day of sensor wear (1-7); Intercept from ANCOVA as agreement rate = 84.59, 91.8% CI 2-sided [82.02 to 87.17] — A group sequential study design was utilized to perform interim analysis. For the final stage, the p-value is 0.041
Statistical Analysis 4: Comparison: Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3) on the Buttock; Test type: Superiority; p < 0.041, ANCOVA; A generalized estimating equation model was used, considering correlation structure of day of sensor wear (1-7); Intercept from ANCOVA as agreement rate = 81.05, 91.8% CI 2-sided [77.58 to 84.53] — A group sequential study design was utilized to perform interim analysis. For the final stage, the p-value is 0.041

ADVERSE EVENTS:
Time Frame: Throughout the course of the study, up to 91 days
Arm/Group | Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) | Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3)
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/142
Serious Adverse Events (participants affected / at risk) | 2/169 | 2/142
Other Adverse Events (participants affected / at risk) | 37/169 | 32/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) (N=169) | Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3) (N=142)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Subjects (Age 18-80) With Diabetes Wearing Guardian™ Sensor (3) (N=169) | Pediatric Subjects (Age 2-17) With Diabetes Wearing Guardian™ Sensor (3) (N=142)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 0 (0)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Medical device site bruise (General disorders) | 1 (1) | 0 (0)
Medical device site haemorrhage (General disorders) | 4 (4) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 1 (1) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 7 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (4) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03966911/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT03966911/SAP_001.pdf